CLINICAL TRIAL: NCT00000714
Title: An Open, Prospective, Multicenter Study of Trimetrexate With Leucovorin Rescue for AIDS Patients With Pneumocystis Carinii Pneumonia (PCP) and Serious Intolerance to Approved Therapies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 039; 11744 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Pneumonia, Pneumocystis Carinii; HIV Infections
Keywords: Trimetrexate; AIDS-Related Opportunistic Infections; Pneumonia, Pneumocystis carinii; Leucovorin; Drug Evaluation; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; Antiprotozoal Agents
MeSH Terms: conditions — Pneumonia, Pneumocystis; HIV Infections; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome | interventions — trimetrexate glucuronate; Leucovorin

INTERVENTIONS:
Drug: Trimetrexate glucuronate
Drug: Leucovorin calcium

SUMMARY:
To determine the safety and effectiveness of an investigational drug therapy (trimetrexate plus leucovorin calcium (TMTX / LCV)) in the treatment of Pneumocystis carinii pneumonia (PCP) in patients who have AIDS, are HIV positive, or are at high risk for HIV infection, and who have suffered severe or life-threatening ill effects from both conventional therapies for PCP. AMENDED: 08/01/90 As of August 31, 1989, 437 patients were enrolled into uncontrolled studies of trimetrexate for PCP:214 in TX 301/ACTG 0=039 (trimetrexate for patients intolerant of approved therapies) and 223 in NS 401 (trimetrexate for patients refractory to approved therapies). The analysis of overall response rate, stringently defined as having received at least 14 days of trimetrexate and being alive at follow-up 1 month after the completion of therapy, reveals 84/159 intolerant patients and 48/160 refractory patients had responded, for rates of 53 percent and 30 percent, respectively. These response rates include all individuals who received at least one dose of trimetrexate. Of the 111 patients who were ventilator-dependent at study entry, 18 completed a course of therapy and were alive a month later, for a response rate of 16 percent. All other ventilated patients died. The most common severe (grades 3 and 4) toxicities were: transaminase elevation (> 5 x normal) in 94 patients, anemia (< 7.9 g/dl) in 109, neutropenia (< 750 cells/mm3) in 58, fever (> 40 C) in 37, and thrombocytopenia (< 50000 platelets/mm3) in 27. Toxicity required discontinuation of therapy in approximately 5 percent of all patients.

Original design: The drugs usually used to treat PCP in AIDS patients, trimethoprim / sulfamethoxazole and pentamidine, have had to be discontinued in many patients because of severe side effects. Currently there are no proven alternatives to these drugs. TMTX was chosen for this trial because it was found to be very active against the PCP organism in laboratory tests. Also TMTX, in combination with LCV, had a high response rate and did not cause severe toxicity in a preliminary trial.

DETAILED DESCRIPTION:
AMENDED: 08/01/90 As of August 31, 1989, 437 patients were enrolled into uncontrolled studies of trimetrexate for PCP:214 in TX 301/ACTG 0=039 (trimetrexate for patients intolerant of approved therapies) and 223 in NS 401 (trimetrexate for patients refractory to approved therapies). The analysis of overall response rate, stringently defined as having received at least 14 days of trimetrexate and being alive at follow-up 1 month after the completion of therapy, reveals 84/159 intolerant patients and 48/160 refractory patients had responded, for rates of 53 percent and 30 percent, respectively. These response rates include all individuals who received at least one dose of trimetrexate. Of the 111 patients who were ventilator-dependent at study entry, 18 completed a course of therapy and were alive a month later, for a response rate of 16 percent. All other ventilated patients died. The most common severe (grades 3 and 4) toxicities were: transaminase elevation (> 5 x normal) in 94 patients, anemia (< 7.9 g/dl) in 109, neutropenia (< 750 cells/mm3) in 58, fever (> 40 C) in 37, and thrombocytopenia (< 50000 platelets/mm3) in 27. Toxicity required discontinuation of therapy in approximately 5 percent of all patients.

Original design: The drugs usually used to treat PCP in AIDS patients, trimethoprim / sulfamethoxazole and pentamidine, have had to be discontinued in many patients because of severe side effects. Currently there are no proven alternatives to these drugs. TMTX was chosen for this trial because it was found to be very active against the PCP organism in laboratory tests. Also TMTX, in combination with LCV, had a high response rate and did not cause severe toxicity in a preliminary trial.

Patients entered in the study are given TMTX for 21 days and LCV for 24 days. Doses are determined by body size. Both drugs are given by intravenous infusion, but LCV may be given orally after the first 10 days. It is essential to ensure that patients receive each and every dose of LCV and that LCV therapy is continued for a full 3 days after TMTX therapy has been completed or discontinued. Doses are adjusted if side effects, such as low white blood cell counts, are too severe. During the 21-day trial, zidovudine (AZT) may not be used, because of possible increased bone marrow toxicity. AZT may be resumed as soon as the administration of TMTX and LCV has been completed.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Noninvestigational therapies as needed.
* Maintenance therapy with investigational triazoles such as itraconazole and SCH 39304.
* High-dose corticosteroids (exceed physiologic replacement doses) including oral prednisone 40 mg bid for 5 days, 40 mg daily for 5 days and then 20 mg daily for the remainder of PCP therapy. Same dose for methylprednisolone.

Concurrent Treatment:

Allowed:

* Any ventilatory support, antihypertensive agents, invasive monitoring, and other necessary medical intervention, according to his/her medical status, personal wishes, and the judgment of his/her physician.

Patients must have:

* HIV seropositivity.
* Diagnosis of Pneumocystis carinii pneumonia (PCP).
* Serious intolerance to trimethoprim / sulfamethoxazole (TMP / SMX) therapy defined as follows:
* Platelets < 50000 platelets/mm3.
* Neutrophil count (polys plus bands) = or < 500 cells/mm3 on at least two occasions = or > 12 hours apart.
* Mucocutaneous reaction - blistering rash, mucosal involvement, generalized maculopapular eruption, or intolerable pruritus.
* Hepatitis demonstrated by transaminase elevation > 5 times the upper limit of normal, or = or > 300 IU if baseline is abnormal.
* Drug fever with daily temperature = or > 103 degrees F beginning after the 5th day of treatment persisting for at least 3 days and not responsive to antipyretic therapy, with no other discernible cause.
* Any other severe or life-threatening adverse reaction to TMP / SMX which, in the investigator's opinion, makes continued or recurrent treatment with TMP / SMX inadvisable as determined on a case-by-case basis.
* Serious intolerance to pentamidine therapy defined as follows:
* Platelets < 50000 platelets/mm3.
* Neutrophil count (polys plus bands) = or < 500 cells/mm3 on at least two occasions = or > 12 hours apart.
* Serum creatinine > 3.0 mg/dl.
* Systolic blood pressure < 90 mm requiring supportive therapy.
* Symptomatic hypoglycemia with blood glucose < 40, or hyperglycemia requiring therapy.
* Pancreatitis with laboratory confirmation (abnormal amylase and/or lipase).
* Any other severe or life-threatening adverse reaction to pentamidine, which, in the investigator's opinion, makes continued or recurrent treatment with pentamidine inadvisable as determined on a case-by-case basis.
* Informed consent by patient or legal guardian.

Prior Medication:

Required:

* Trimethoprim / sulfamethoxazole and pentamidine therapies.

Prior Medication:

Allowed:

* Myelosuppressive or nephrotoxic agents including zidovudine.

History of high-risk behavior for HIV infection - homosexual or bisexual men, intravenous drug abusers, recipients of HIV-infected blood products, or sexual partners of persons in these groups may be admitted without proof of HIV infection.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* History of Type I hypersensitivity (i.e., urticaria, angioedema, or anaphylaxis), exfoliative dermatitis, or other life-threatening reactions due to trimetrexate.
* Patients with a less severe adverse reaction may be enrolled if, in the opinion of the investigator, these adverse effects do not prohibit rechallenge with the drug.

Concurrent Medication:

Excluded:

* Myelosuppressive or nephrotoxic agents including zidovudine and ganciclovir.
* Investigational therapies.

Patients with the following are excluded:

* History of Type I hypersensitivity (i.e., urticaria, angioedema, or anaphylaxis), exfoliative dermatitis, or other life-threatening reactions due to trimetrexate.
* Patients with a less severe adverse reaction may be enrolled if, in the opinion of the investigator, these adverse effects do not prohibit rechallenge with the drug.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Study Completion 2004-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Feinberg J, Study Chair
Locations (21):
- United States (21):
  - Univ of Miami School of Medicine, Miami, Florida
  - Northwestern Univ Med School, Chicago, Illinois
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Tulane Univ School of Medicine, New Orleans, Louisiana
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Beth Israel Deaconess - West Campus, Boston, Massachusetts
  - Univ of Massachusetts Med Ctr, Worcester, Massachusetts
  - Warner-Lambert Parke-Davis, Morris Plains, New Jersey
  - SUNY / Erie County Med Ctr at Buffalo, Buffalo, New York
  - City Hosp Ctr at Elmhurst / Mount Sinai Hosp, Elmhurst, New York
  - Beth Israel Med Ctr, New York, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - SUNY - Stony Brook, Stony Brook, New York
  - Bronx Municipal Hosp Ctr/Jacobi Med Ctr, The Bronx, New York
  - Montefiore Med Ctr / Bronx Municipal Hosp, The Bronx, New York
  - Duke Univ Med Ctr, Durham, North Carolina
  - Case Western Reserve Univ, Cleveland, Ohio
  - Julio Arroyo, West Columbia, South Carolina
  - Univ of Washington, Seattle, Washington

REFERENCES:
- [Background] Katz D, Feinberg J, Myers M, Gubish E, Hoth D. Providing access to promising investigational drugs for AIDS: A management model for "treatment INDs". Int Conf AIDS. 1989 Jun 4-9;5:855 (abstract no TEP51)
- [Background] Feinberg J, Katz D, McDermott C, Myers M, Hoth D. Trimetrexate (TMTX) salvage therapy of PCP in AIDS patients without any therapeutic options: interim results of the 1st AIDS "treatment IND" protocol. Int Conf AIDS. 1989 Jun 4-9;5:201 (abstract no TBO28)